CLINICAL TRIAL: NCT02786225
Title: Interprofessional Perinatal Consults to Improve Communication Quality, Satisfaction, and Team Cohesion: A Randomized Trial of the Collaboration for Antepartum Risk Evaluation (CARE) Model
Brief Title: Collaboration for Antepartum Risk Evaluation
Acronym: CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Julia Phillippi, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 160523
Record Dates: First submitted 2016-05-18; First posted 2016-05-30 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Prenatal Care; Maternal-child Health Services; Maternal Health Services; Perinatal Care; Midwifery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Collaborative Care (Experimental): Intervention Group: Women (n=118) will be seen one time, simultaneously by a Vanderbilt University Medical Center (VUMC) perinatologist and a Vanderbilt University School of Nursing (VUSN) nurse-midwife (the CARE visit). During the CARE visit, the nurse-midwife and perinatologist will complete the CARE checklist The checklist will be signed by the woman and providers and scanned into the medical record. Following the CARE visit, women will return to midwifery care or be referred to perinatology depending on their needs, remaining in the study. Women returning to the midwifery practice will see a primary midwife for the remainder of care.
  Interventions: Behavioral: Collaborative Care
- Comparison Care- Usual Care + primary midwife (Active Comparator): Comparison Group: Usual care enhanced with primary midwife. Women in the comparison group (n=118) will receive the standard individual consult visit with a perinatologist and then, if they return to midwifery care, have one consistent midwife (primary midwife) for the majority of remaining prenatal care.
  Interventions: Behavioral: Comparison Care- Usual Care + primary midwife

INTERVENTIONS:
Behavioral: Collaborative Care — Intervention Group: Women (n=118) will be seen one time, simultaneously by a VUMC perinatologist and a VUSN nurse-midwife (the CARE visit). During the CARE visit, the nurse-midwife and perinatologist will complete the CARE checklist The checklist will be signed by the woman and providers and scanned into the medical record. Following the CARE visit, women will return to midwifery care or be referred to perinatology depending on their needs, remaining in the study. Women returning to the midwifery practice will see a primary midwife for the remainder of care.
  Arms: Collaborative Care
Behavioral: Comparison Care- Usual Care + primary midwife — Comparison Group: Usual care enhanced with primary midwife. Women in the comparison group (n=118) will receive the standard individual consult visit with a perinatologist and then, if they return to midwifery care, have one consistent midwife (primary midwife) for the majority of remaining prenatal care.
  Arms: Comparison Care- Usual Care + primary midwife

SUMMARY:
Perinatal outcomes in the US rank behind most other developed countries even though women in the US utilize more maternity services. Current approaches to consultation and collaboration among perinatal care providers, including nurse-midwives, obstetricians, and perinatologists, fragment care resulting in communication errors and maternal dissatisfaction. The CARE study will test an innovative interdisciplinary consult visit to improve communication, teamwork, maternal satisfaction, and perinatal outcomes.

DETAILED DESCRIPTION:
Perinatal outcomes in the United States rank below many other developed countries. National organizations, such as the American College of Obstetricians and Gynecologists, have called for women to utilize the level and provider of maternity services that meet their personal and medical needs. This leveled approach to care requires consultation and collaboration among providers to ensure women receive appropriate services. While national and international organizations have called for team-based maternity care, current models can fragment services, increasing the risk of communication errors. Women can feel disenfranchised by models that do not meet their needs and opt out of beneficial services altogether.

Currently, there is not evidence on effective interdisciplinary models of maternity care. The Collaboration for Antepartum Risk Evaluation (CARE) study will use a randomized design to systematically test the effect of interdisciplinary consults on women and providers. The two aims of the study are: (1) evaluate the effect of collaborative vs individual consults on participant outcomes including communication quality (using the Communication Assessment Tool, team version), maternal satisfaction (using a modified Satisfaction with Prenatal Care measure), semi-structured interviews, adherence to the developed plan of care, and perinatal outcomes; (2) evaluate the effect of the CARE clinic on providers using the Communication Assessment Tool- team version, the Agency for Healthcare Research and Quality (AHRQ) Team Strategies and Tools to Enhance Performance and Patient Safety (TeamSTEPPS) questionnaire, and semi-structured interviews.

The CARE study will provide valuable information on effective models for patient-centered maternity care. The AHRQ K08 will allow Dr. Philippi to implement the CARE study and facilitate her growth into a national leader in midwifery and health services research.

ELIGIBILITY:
Inclusion Criteria:

* Adult pregnant women receiving prenatal care at the VUSN Nurse-Midwifery Faculty Practice.
* Gestational age of pregnancy 4-40 weeks
* Needs a consultation with perinatologist for one of the following reasons:

Prior pregnancy with congenital abnormality History of fetal demise >20 weeks History of preterm labor in previous pregnancy Current maternal drug or alcohol abuse Controlled maternal condition (e.g. thyroid disorder) Mild abnormality of fetus or placenta on ultrasound Idiopathic thrombocytopenia in pregnancy

* Can attend the collaborative care clinic

Exclusion Criteria:

* Unable to give consent for research participation - including age < 18 or impaired mental function
* Urgent medical condition requiring immediate assessment including: ectopic pregnancy or vaginal bleeding
* Medical conditions outside of scope of VUSN midwifery guidelines including:

Chronic maternal conditions requiring specialist involvement including: HIV, epilepsy, uncontrolled asthma, and liver, renal, cardiac disease.

Multiple gestation > 2 previous cesarean births Rh isoimmunization Incompetent cervix Major fetal or placenta abnormalities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2016-07; Primary Completion 2020-10 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Communication Assessment Tool (CAT)-Team survey | 2 weeks after intervention/comparison visit
  The CAT, developed by Makoul et al., assesses views of provider communication via 14 Likert responses ranging from 1= 'poor' to 5= 'excellent.
Satisfaction with Prenatal Care (SPC) scale | 2 weeks after intervention/comparison visit
  The SPC scale assesses patient satisfaction with prenatal care
Communication Assessment Tool (CAT)-Team survey - following birth | Within 2 weeks after patient gives birth
  The CAT, developed by Makoul et al., assesses views of provider communication via 14 Likert responses ranging from 1= 'poor' to 5= 'excellent.
Satisfaction with Prenatal Care (SPC) scale - following birth | Within 2 weeks after patient gives birth
  The SPC scale assesses patient satisfaction with prenatal care

SECONDARY OUTCOMES:
Smoking at 1st prenatal visit | 1 week after the patient gives birth
For smokers, number of cigarettes per day | 1 week after the patient gives birth
  Number of cigarettes per day
Location of birth | 1 week after patient gives birth
  Location where the mother gave birth - Vanderbilt / Other hospital, Birth center, Home, En Route
Provider at admission to labor and delivery | 1 week after patient gives birth
  Medical care provider at the time of admission in labor
Patient & provider adherence to checklist plan | 1 week after patient gives birth
  Congruence between the anticipated plan of care at the time of the intervention/comparison visit and what occurred at the time of birth
Gestational age at birth | 1 week after patient gives birth
  the gestational age of the baby at the time of birth - in weeks+days
Infant birth weight | 1 week after patient gives birth
  Infant birth weight in grams as collected within 4 hours of birth
Mode of birth | 1 week after patient gives birth
  Number of women giving birth via 1 of 4 methods: vaginal/assisted vaginal/cesarean after labor/planned cesarean
Trial of labor after cesarean | 1 week after the mother gives birth
  Whether the woman was attempting a trial of labor after a previous cesarean birth
Vaginal birth after cesarean | 1 week after patient gives birth
  Whether the woman gave birth vaginally with this infant after she had a previous cesarean birth.
Complications at birth | 1 week after patient gives birth
  The presence of any adverse outcomes during pregnancy, birth, postpartum, including details
Breastfeeding at birth | 1 week after patient gives birth
  Breastmilk feeding of the infant at the time of birth
Breastfeeding at discharge | 1 week after patient gives birth
  Breastmilk feeding of the infant at the time of discharge.
Hospital stay postpartum | 1 week after patient gives birth
  Lengths of postpartum hospital stay in calendar days
Generalized Anxiety Disorder 7-item scale (GAD-7) | 2 weeks after intervention/comparison visit
  Measure of anxiety level. Scale can range from 0-21 with higher scores representing greater anxiety.
Generalized Anxiety Disorder 7-item scale (GAD-7) | Within 2 weeks after patient gives birth
  Measure of anxiety level. Scale can range from 0-21 with higher scores representing greater anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Phillippi, PhD, Principal Investigator — Vanderbilt School of Nursing
Locations (1):
- Vanderbilt School of Nursing, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share deindentified data after submission of the Data Use Agreement
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Will share deindentified data after submission of the Data Use Agreement
Access Criteria: To be determined

REFERENCES:
- [Derived] Phillippi JC, Doersam JK, Neal JL, Roumie CL. Electronic Informed Consent to Facilitate Recruitment of Pregnant Women Into Research. J Obstet Gynecol Neonatal Nurs. 2018 Jul;47(4):529-534. doi: 10.1016/j.jogn.2018.04.134. PMID 29758172